CLINICAL TRIAL: NCT02555943
Title: Direct Antiviral Agents for the Treatment of Chronic HCV/HBV Co-infection Patients
Brief Title: DAAs Treatment for Chronic HCV/HBV Co-infection Patients(DASCO)
Acronym: DASCO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, George Lau, Director, Humanity and Health Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&H_DASCO
Record Dates: First submitted 2015-09-20; First posted 2015-09-22 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis C Infection; HBV Coinfection; Hepatitis B Reactivation
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination; Sofosbuvir; ledipasvir; daclatasvir; Viekira Pak; entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic/Early anti-HBV treatment (Active Comparator): HCV/HBV co-infection patients in this arm will receive nucleos(t)ides analog (Entecavir or Tenofovir disoproxil fumarate) for the treatment of hepatitis B infection before or at the commencement of direct anti-HCV treatment using DAAs (Ledipasvir/Sofosbuvir; or Sofosbuvir and Daclatasvir, or Ombitasvir, Paritaprevir, Ritonavir, Dasabuvir; or Sofosbuvir+Ribavirin).
  .
  Interventions: Drug: Ledipasvir/Sofosbuvir; Drug: Sofosbuvir and Daclatasvir; Drug: Ombitasvir, Paritaprevir, Ritonavir, Dasabuvir; Drug: Entecavir; Drug: Tenofovir disoproxil
- Deferred anti-HBV treatment (Experimental): HCV/HBV co-infection patients in this arm will receive nucleos(t)ides analog (Entecavir or Tenofovir disoproxil fumarate) for the treatment of hepatitis B infection when HBV viral breakthrough occurred during anti-HCV treatment using DAAs (Ledipasvir/Sofosbuvir; or Sofosbuvir and Daclatasvir, or Ombitasvir, Paritaprevir, Ritonavir, Dasabuvir; or Sofosbuvir+Ribavirin).
  Interventions: Drug: Ledipasvir/Sofosbuvir; Drug: Sofosbuvir and Daclatasvir; Drug: Ombitasvir, Paritaprevir, Ritonavir, Dasabuvir; Drug: Entecavir; Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Ledipasvir/Sofosbuvir — Oral direct anti-HCV agent. Ledipasvir/Sofosbuvir(LDV/SOF) 400mg/90mg fixed-dose combination(FDC) tablet, administered orally once daily.
  Other Names: Harvoni®; GS-7977; GS-5885
Drug: Sofosbuvir and Daclatasvir — TWO oral direct anti-HCV agent: Sofosbuvir(SOF), 400mg tablet administered orally once daily. Daclatavir(DCV), 60mg tablet administered orally once daily.
  Other Names: Sovaldi®, GS-7977; Daklinza®,BMS-790052
Drug: Ombitasvir, Paritaprevir, Ritonavir, Dasabuvir — VIEKIRA PAK includes ombitasvir, a hepatitis C virus NS5A inhibitor, paritaprevir, a hepatitis C virus NS3/4A protease inhibitor, ritonavir, a CYP3A inhibitor and dasabuvir, a hepatitis C virus non-nucleoside NS5B palm polymerase inhibitor.
  Other Names: VIEKIRA PAK™
Drug: Entecavir — Nucleoside-inhibitor-treatment-naïve with compensated liver disease (greater than or equal to 16 years old): 0.5 mg once daily.
  Other Names: BARACLUDE®
Drug: Tenofovir disoproxil — VIREAD is indicated for the treatment of chronic hepatitis B in adults and pediatric patients 12 years of age and older.
  Other Names: VIREAD®

SUMMARY:
This is a prospective study to determine the incidence, morbidity, mortality and predisposing factors for the reactivation of hepatitis B virus replication during direct anti-HCV treatment of HCV/HBV co-infection patients.

DETAILED DESCRIPTION:
Patients who receive direct-acting anti-HCV treatment will be prospectively studied during 2-year period. All patients have HCV/HBV co-infection.

The inclusion/exclusion criteria and the follow up plan will be listed in following part.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA positive,
* HBsAg positive with detectable or undetectable HBV DNA,
* Receiving pan oral direct-acting anti-HCV regimen

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner;
* HIV infection;
* Hematologic or biochemical parameters at Screening outside the protocol- specified requirements;
* Active or recent history (≤ 1 year) of drug or alcohol abuse;
* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who experience virological breakthrough | From the commencement of DAAs treatment to 12 weeks post DAAs treatment
  Virological breakthrough is defined as 1 logIU/ml increase during and/or post DAAs treatment for the baseline or nadir.
Proportion of participants who experience virological rebound | From the commencement of DAAs treatment to 12 weeks post DAAs treatment
  Virological rebound is defined as 2 logIU/ml increase during and/or post DAAs treatment for the baseline or nadir.

SECONDARY OUTCOMES:
Proportion of participant who experience biochemical rebound | From the commencement of DAAs treatment to 12 weeks post DAAs treatment
  Biochemical rebound is defined as

OTHER OUTCOMES:
Proportion of participant who experience liver failure | From the commencement of DAAs treatment to 12 weeks post DAAs treatment
  Diagnosis of liver failure

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, M.D., Principal Investigator — Humanity and Health GI and Liver Centre
Locations (1):
- Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong, China